CLINICAL TRIAL: NCT04316312
Title: The Inspiratory Muscle Activation Pattern and Training Efficacy in Patients With Chronic Obstructive Pulmonary Disease After Acute Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201912165RINB
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory muscle training group (Experimental)
  Interventions: Device: Threshold inspiratory muscle trainer

INTERVENTIONS:
Device: Threshold inspiratory muscle trainer — Threshold inspiratory muscle trainer will be set between 15% to 30% of maximal inspiratory pressure.

SUMMARY:
The purpose of this study is to assess the activation patterns of diaphragm and sternocleidomastoid (SCM) muscle during different loaded inspiratory muscle performance in patients with COPD after acute exacerbation. Null hypothesis (H0): There is no significant difference between activation pattern of diaphragm and SCM muscle during different loaded inspiratory muscle performance in patients with COPD after acute exacerbation. Alternative hypothesis (H1): There is significant difference between activation pattern of diaphragm and SCM muscle during different loaded inspiratory muscle performance in patients with COPD after acute exacerbation.

DETAILED DESCRIPTION:
The prevalence of chronic obstructive pulmonary disease (COPD) is 11.7% around the world, and it is expected to rise over the next 30 years. In Taiwan, COPD is estimated as the seventh leading cause of death in 2016, and has been gradually increasing in the past decades. COPD has been long considered to be a disease state characterized by airflow limitation that are not fully reversible, leading to abnormalities in control of breathing, worsening of respiratory mechanics and pulmonary function. However, COPD is no longer considered to affect only the lungs and airways, but also the rest of the body including decreases in respiratory and limb-muscle mass and function. When acute exacerbation occurs, lung function decreases rapidly. According to the previous studies, inspiratory muscle training (IMT), can improve the strength and endurance of the diaphragm, reduce dyspnea and breathing pattern, thus increasing the capacity of activities tolerance in patients with COPD. Although more and more studies are focus on diaphragm weakness and the effect of IMT in patients with COPD, the efficacy and intensity of IMT in patients with COPD is still controversial and the clinical use is limited. Whether increases intensity during IMT would lead to improvements in contraction pattern of respiratory muscle remained unclear. Therefore, the purpose of this study is to assess the activation patterns of diaphragm and sternocleidomastoid (SCM) muscle during different loaded inspiratory muscle performance in patients with COPD after acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years old
* has been diagnosis of chronic obstructive pulmonary disease and experienced at least 2 times of acute exacerbation in recent 6 months
* can cooperate with the measurements of this study

Exclusion Criteria:

* any clinical diagnosis that will influence the measurement, including any history of neuromyopathy
* angina, acute myocardial infarction in the previous one month
* pregnancy
* participated in inspiratory muscle training program in the previous three months
* any psychiatric or cognitive disorders, for example: Mini-Mental State Examination (MMSE) < 24, that will disturb the communication and cooperation of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Diaphragm and Sternocleidomastoid muscle activation | through the completion of the maximal inspiratory pressure test and loaded inspiratory muscle test condition; totally it would take about 3 minutes
  The surface electromyography (EMG) signal was analyzed in the time domain, calculating root mean square (RMS) amplitude with a time constant of 30 mini seconds. A 1.5 seconds window of diaphragm and SCM muscle signals at peak pressure during maximal inspiratory pressure test were obtained and calculated as maximal effort. Diaphragm and SCM activation were calculated using mean RMS values of each threshold loaded breathing test, and then normalized to maximal effort (%EMGDia and %EMGSCM).

SECONDARY OUTCOMES:
The mean median frequency of diaphragm and sternocleidomastoid muscle | In one minute after the completion of the loaded inspiratory muscle test condition
  The power spectrum is divided into two equal areas of the frequency value by median frequency to exam muscle fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, PhD, Study Chair — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy of National Taiwan University, Taipei, Zhongzheng Dist, Taiwan